CLINICAL TRIAL: NCT07217574
Title: Care Coordination and Communication Program in Oncology for Tribal Health Systems (C3PO)
Brief Title: Program in Oncology for Tribal Health Systems.
Status: Recruiting | Type: Observational
Sponsor: University of Oklahoma (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: Tribal Health C3PO; U19MD020537 (NIH)
Record Dates: First submitted 2025-09-26; First posted 2025-10-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Patient Outcomes
Keywords: American Indian (AI); American Native (AN)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Open Pilot Study: During the open pilot study, which will take place over a 3-month period, up to 15 patients will be enrolled to receive the C3PO intervention. At the conclusion of this period, exit interviews will be conducted to gather feedback on the implementation of the intervention. The primary objective of this phase is to assess the strengths and weaknesses of the intervention in order to inform potential improvements before advancing to the next phase of the study
  Interventions: Other: C3PO
- C3PO Intervention: In Phase II of the study, patients will be randomized 1:1 by site and cancer type to either the C3PO intervention group or the usual care group. Those assigned to the C3PO arm will receive navigation services at SCC, along side collaborative care meetings (C3PO). These meetings, held without the patient present, will focus on discussing the patient's overall needs, such as potential adverse effects of cancer treatment, the impact of co-morbid conditions, etc,.
  Interventions: Other: C3PO
- Usual Care: Patients randomized to the usual care group will receive navigation services only and will not participate in the C3PO intervention during the initial 6 months. However, after this 6-month period, they will become eligible to receive the C3PO intervention, following the same process as the initial intervention group.
  Interventions: Other: C3PO

INTERVENTIONS:
Other: C3PO — Participants assigned to C3PO will receive usual navigation services with a Native American Navigator (NAN) at the SCC but will begin having their clinical care and social needs discussed during monthly collaborative care meetings. For the Open Pilot, this will include all participants (no randomization or usual care group). The collaborative care coordinator will meet with the participant virtually or in-person before and after collaborative care meetings as they are available and as needs arise.

SUMMARY:
This clinical trial aims to develop and implement more navigation assistance programs tailored specifically for Native American cancer patients, addressing the current lack of available support. The goal is to improve communication barriers within the healthcare system by fostering a collaborative approach between the Stephenson Cancer Center (SCC) and tribally operated healthcare systems (ITU). Through this partnership, the trial seeks to enhance patient outcomes by providing culturally sensitive, coordinated care.

DETAILED DESCRIPTION:
This study aims to evaluate the impact of collaborative care meetings (CCM) on patient-reported outcomes through a two-phase approach including Native American patients with cancer. Phase I is a 3-month pilot with up to 15 patients completing baseline assessments, monthly surveys, and exit interviews. Phase II is a randomized controlled trial (RCT) comparing the Care Coordination and Communication Program in Oncology for Tribal Health Systems (C3PO) intervention to usual care (standard Native American navigation services), with all participants accessing the C3PO intervention after 6 months. C3PO meetings will address treatment side effects, comorbidities, approvals for referred care, and barriers such as transportation or financial hardship.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be at least 18 years of age, within eight weeks of newly diagnosed cancer confirmed by pathology/imaging, navigated through the NANP at SCC and have verbal fluency in English.

Exclusion Criteria:

* Participants in the Phase 1 open pilot will not be eligible for the Phase 2 RCT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include all race and ethnic groups for staff interviews. Patient interviews and surveys will be restricted to American Indian/American Native patients.
Sampling Method: Probability Sample
Enrollment: 187 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Perceptions of Cancer Care Coordination Needs | 1 year
  All participants will complete the Patient Satisfaction with Cancer Care (PSCC) at baseline and monthly during the study duration.

SECONDARY OUTCOMES:
Number of Missed Visits | 2 years
  Completed and all missed visits will be recorded in SCC's appointment database, which will be queried via the institutional software. The NANP cohort will be run through this query monthly to identify missed oncology visits, and the information will be entered into the NANP database. The proportion of missed visits for all navigated patients will be tallied monthly. Types of missed visits include no-show, canceled by SCC, rescheduled by pt, other, and unknown.
Time from Diagnosis to Initial Treatment | 3 years
  Using the EHR, in partnership with the OU Clinical Research Data Warehouse, we will calculate the average number of days from date of diagnosis to date of first treatment for existing and newly navigated patients.

OTHER OUTCOMES:
Treatment Interruptions | 4 year
  For treatment alignment, we will assess for alignment between treatment recommended and fitness (measured as met vs. not met) and alignment between treatment received and recommended (measured as met vs. not met). Alignment between fitness and treatment will be assessed using National Comprehensive Cancer Network (NCCN) recommendations and agreed upon by the physicians.
Treatment Intensity | 4 year
  For treatment intensity, we will evaluate relative dose intensity defined as the ratio of the total dose of treatment actually delivered relative to the standard treatment dose. Doses of treatments will be captured for initial treatment and characterized as full dose vs. dose reduced. For complications, the treatment modifications (dose reductions and delays) will be abstracted for medical therapies.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Janitz, Ph.D., Principal Investigator — University of Oklahoma Stephenson Cancer Center
Locations (1):
- OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No